CLINICAL TRIAL: NCT06718946
Title: A Phase I Clinical Study on the Safety and Efficacy of Intravenous Administration of IDOV-SAFETM in the Treatment of Advanced Solid Tumors
Brief Title: Study on the Safety and Efficacy of Intravenous Administration of IDOV-SAFETM in the Treatment of Advanced Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Hongxia Wang, Chief of Internal Medicine, Fudan University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LY001-F001
Record Dates: First submitted 2024-09-11; First posted 2024-12-05 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-12

CONDITIONS: Advanced Malignant Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oncolytic Virus injection(IDOV-SAFETM) (Experimental): Intravenous administration of IDOV-SAFETM every 3 weeks for patients with advanced solid tumors.
  Dose cohorts: 3x10^8 PFU、7x10^8 PFU 、1x10^9 PFU、3x10^9 PFU、7x10^9 PFU 、1x10^10 PFU and 3x10^10 PFU
  Interventions: Biological: IDOV-SAFE

INTERVENTIONS:
Biological: IDOV-SAFE — Intravenous administration of oncolytic virus every 3 weeks until tumor progression

SUMMARY:
This is an open-label, dose escalation, phase I study to evaluate safety tolerability, MTD, pharmacokinetic profile, immunogenicity, and pharmacodynamic profile of Intravenous Administration of IDOV-SAFETM in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The therapeutic dose for mice was 1x10^8 PFU, and the maximum starting dose for humans was 2.67x10^9 PFU based on the Guidelines for Estimating the Maximum Recommended Starting Dose for the First Clinical Trial of Healthy Adult Volunteers.

Dose escalation phase:

At this stage, the investigators plan to enroll about 17-32 patients with advanced solid tumors who have failed standard treatment in China to conduct intravenous administration of IDOV-SAFETM.

This phase includes seven dose groups of 3x10^8 PFU, 7x10^8 PFU, 1x10^9 PFU, 3x10^9 PFU, 7x10^9 PFU, 1x10^10 PFU and 3x10^10 PFU. The first dose group includes 1 subject. If the subject does not develop DLT, The next dose group should be opened for treatment. If this subject develops DLT, the dose group and all subsequent dose groups should be increased by the conventional "3+3" method. For the dose group with "3+3" dose increment, 3 to 6 subjects were enrolled in each group. Each patient received intravenous administration on the first day, with a course of 21 days. The follow-up investigator decided whether to continue the second (D22) course of administration according to the comprehensive assessment of the subjects' conditions; All subjects in each dose group may be incremented to the next dose group after completing a safety assessment 21 days after the first dose.

The dose escalation or setting may be adjusted as determined by the Safety Committee (SMC).

Dose expansion phase:

In the dose expansion phase, the previous dose or an intermediate dose of MTD and the clinical dosage to be used later were selected to carry out the expansion experiment, and 6 subjects were expanded. Each patient received intravenous administration on the first day, and the treatment course was 21 days. The follow-up researchers decided whether to continue the administration of the second course (D22) according to the comprehensive evaluation of the subjects' conditions. Each patient was treated for at least one course of treatment (22 days).

Based on the preliminary clinical trial data, the number of injections and the interval time of administration can be adjusted during the dose expansion phase after the decision of the Safety Committee (SMC).

Duration of administration:

In both phases, safety and efficacy were evaluated 42 days after initial dosing. If CT evaluation suspects false progression, puncture and pathology examination are required.

After SMC's decision, it is determined that the benefits of continued treatment outweigh the risks of the subject, and if the subject wishes to continue treatment, the subject may continue to receive the experimental drug. The specific course of treatment will be determined by the SMC based on preliminary clinical trial data.

The safety and efficacy of the investigational drug will be evaluated periodically during continued dosing, and the risk and benefit of continuing treatment will be determined by the SMC. If benefit > risk is no longer satisfied, the long-term safety and survival follow-up period is entered.

Long-term safety and survival follow-up:

Adverse events occurring throughout the study from the first dosing of each subject in both phases will be collected, and long-term safety and survival follow-up will continue up to 2 years after the last dosing (telephone survival follow-up every 8 weeks from the last dosing until the patient meets end-of-treatment criteria or end-of-survival follow-up date, whichever arrives first).

ELIGIBILITY:
Inclusion Criteria:

1. Age: from 18 to 75 years old.
2. At the time of screening, the patient had at least one measurable target lesion.
3. Patients with advanced solid tumors who have failed standard therapy during screening.
4. When screening, the ECOG score of physical strength score is 0 or 1.
5. Life expectancy assessed by the investigator at the time of screening was ≥3 months.
6. Subject has qualified organ function at baseline:

   a) Bone marrow function (no growth factor support therapy or component transfusion within 14 days prior to screening) : i. Neutrophil absolute value (ANC) ≥1.5×10^9/L; ii. Hemoglobin (HB) ≥90g/L; iii. Platelet count (PLT) ≥75×10^9/L; b) Liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times the upper limit of normal (ULN), total bilirubin (TBIL) ≤1.5 times ULN (ALT and AST≤5 times ULN, TBIL≤3 times ULN for liver metastasis or hepatocellular carcinoma); c) Renal function: serum creatinine ≤ULN or creatinine clearance ≥80mL/min;
7. Fertile female subjects must have negative blood beta-HCG test results within 7 days prior to enrollment.
8. Subjects must agree to use highly effective contraception for at least 90 days from the start of the ICF to the end of the study.
9. Be fully informed of this study and voluntarily sign ICF.

Exclusion Criteria:

1. Asymptomatic brain metastases such as untreated ones at the time of screening; Subjects with symptomatic central nervous system (CNS) metastatic or cancerous meningitis; Or there was other evidence of uncontrolled central nervous system or meningeal metastases in subjects who were judged by the investigator to be unsuitable for enrollment.
2. Prior to enrollment, there was severe chronic or active infection: active hepatitis B (HbsAg positive, HBV DNA test value greater than the upper limit of normal); Active hepatitis C (those with positive anti-HCV antibodies are further tested positive for HCV RNA); A known history of immunodeficiency virus (HIV) disease or a positive HIV antibody test; Other conditions requiring systemic anti-infective treatment in the 4 weeks prior to initial use of the investigational drug include, but are not limited to, hospitalization for infectious complications, bacteremia, severe pneumonia, or active tuberculosis.
3. At the time of screening, patients had a history of active autoimmune diseases such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc., or were receiving long-term systemic steroids (prednisone >10mg/ day or equivalent doses of the same drug) or any other form of immunosuppressant therapy within 4 weeks prior to the first use of the study drug.
4. Patients with received allogeneic tissue or solid organ transplantation.
5. There is evidence of clinically significant immunodeficiency, such as primary immunodeficiency status, such as severe combined immunodeficiency disease (SCID); Combined with opportunistic infections.
6. Anticoagulants or antiplatelet drugs should be used before injection and should not be interrupted, including: aspirin should not be stopped within 7 days before injection; Coumarin that cannot be stopped within 7 days prior to injection; Direct thrombin inhibitors (such as dabigatrun) or direct factor Xa inhibitors (such as rivaroxaban, apixaban, and neperoxaban) that cannot be discontinued within 4 days prior to injection; Low molecular weight heparin (LMWH) should not be stopped within 24 hours before injection, and ordinary heparin (UFH) should not be stopped more than 4 hours before injection.
7. Patients with a history of severe cardiovascular and cerebrovascular disease, including but not limited to: congestive heart failure ≥II heart function grade of the New York Heart Association (NYHA); Left ventricular ejection fraction (LVEF) <50%; QT interval (QTcF) >470ms as corrected by the Fridericia method or prolonged QT interval syndrome; Acute coronary syndrome, aortic dissection, severe arrhythmia, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events occurred within 6 months before first administration; The presence of uncontrolled hypertension (systolic blood pressure >140mmHg or diastolic blood pressure >90mmHg). Subjects with a history of hypertension are admitted to the study if their blood pressure is controlled and maintained below this standard with antihypertensive therapy.
8. Patients with received treatment with other methods, including but not limited to chemotherapy, radiotherapy, biotherapy, endocrine therapy, immunotherapy, etc., within 4 weeks prior to the first use of the investigational drug.
9. Other diseases or abnormalities assessed by the investigator as unsuitable for participation in the study.
10. Vaccination against smallpox or monkeypox within 10 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | up to 3 weeks
  Dose-limiting toxicity is defined as an adverse event that is considered to be drug-related and meets one of the Protocol definitions
MTD | up to 3 weeks
  To explore the maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
Levels of viral DNA in blood | up to 3 days
  Peripheral blood was collected for viral DNA and live viral load measurement
Tumor markers | through study completion, an average of 1 year
  Blood samples are used to determine tumor markers.
T cell subsets | through study completion, an average of 1 year
  Analysis 1: Reactivation of memory T cells; Analysis 2: Multifunctional recovery of exhausted T cells.
Objective response rate | through study completion, an average of 1 year
  The sum of the proportion of subjects with Complete response or Partial response
Disease control rate | through study completion, an average of 1 year
  The sum of the proportion of subjects with Complete response 、Partial response or Stable disease
Progression Free Survival | through study completion, an average of 1 year
  The time, measured in days, from the date of first treatment to disease progression or death from any cause. Disease progression and death were measured in terms of preoccurrence. Progression included radiographic progression or clinical progression as assessed by the investigator.
Overall Survival | 2 years
  The time from the date of first treatment to death from any cause, measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Wang, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China